CLINICAL TRIAL: NCT04325321
Title: Heterogeneity and Predictors of Stress Reactivity in Takotsubo Syndrome
Brief Title: The Broken Heart Study II (BHS-II)
Acronym: BHS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Elena Salmoirago-Blotcher, Senior Research Scientist, Associated Professor of Medicine, The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01HL149672 (NIH); R01HL149672 (NIH)
Record Dates: First submitted 2020-03-23; First posted 2020-03-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Takotsubo Cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress reactivity (Other): Stress reactivity test
  Interventions: Other: Stress reactivity test

INTERVENTIONS:
Other: Stress reactivity test — The protocol consists of Resting Baseline (BL), Emotion Recall (ER), followed by a Recovery Phase (RP). Heart rate and blood pressure are measured at baseline and then every 5 minutes during ER and RP.
  Resting Baseline (BL - 10 min). The participant is instructed to rest quietly.
  Emotion Recall (ER - 5-10 min). The participant is instructed to think about the incident associated with the onset of their cardiac event and bring to mind details of the incident. When the participants have the incident clearly in mind, they are instructed to relate the incident and their experience out loud; frequent questions to re-elicit the emotion are asked.
  Recovery Phase (RP - 20 min). Upon completion of RP, the catheter is removed and participants are de-instrumented. Blood samples for plasma catecholamines, assessments of heart rate variability, and echocardiograms are performed 10-min into BL, 10-min into ER, and 18 minutes into RP.

SUMMARY:
The goals of this study are as follows:

1. To rigorously establish and characterize heterogeneity in the pathophysiology of Takotsubo Syndrome (TS).
2. To rigorously test the contribution of TS triggering events and mental stress responsiveness to 1-year prognosis after TS event.

DETAILED DESCRIPTION:
Newly admitted patients with a validated diagnosis of Takotsubo Syndrome (TS; n=106) will be enrolled from 3 large medical centers in the Providence, Rhode Island area. Between 2 and 4 weeks after discharge, clinically stable patients will undergo an in-person comprehensive interview to identify the events proximal to the onset of TS symptoms, complete a battery of psychosocial questionnaires and undergo a validated laboratory stress protocol. Baseline and reactive changes in measures of autonomic nervous system activity (epinephrine and norepinephrine - primary outcome), and in the secondary outcomes of cardiac vagal control and left ventricular function (ejection fraction; regional and global longitudinal strain assessed with speckle tracking echocardiography) will be assessed. Echocardiographic evaluations will be repeated 12 months thereafter together with information on major adverse cerebrovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18
* A new diagnosis of takotsubo syndrome fulfilling Mayo Clinic criteria
* Ability to understand and speak English

Exclusion Criteria:

* Inability or unwillingness to give informed consent
* Severe cognitive impairment
* Uncontrolled hypertension
* Acute psychosis
* High suicidal risk
* Pregnancy
* Poor echocardiographic window
* Conditions that would interfere with adherence to study requirements (e.g., ongoing alcohol or substance abuse)
* If the participant is clinically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Mean change (in pg/mL) in plasma epinephrine levels | Up to 4 weeks
  Blood samples for plasma epinephrine are collected 10-min into Baseline, 10-min into Emotion Recall, and 18 minutes into Recovery Phase. Change will be calculated by subtracting Baseline epinephrine levels from Emotion Recall levels.
Mean change (in pg/mL) in plasma norepinephrine levels | Up to 4 weeks
  Blood samples for plasma norepinephrine are collected 10-min into Baseline, 10-min into Emotion Recall, and 18 minutes into Recovery Phase. Change will be calculated by subtracting Baseline epinephrine levels from Emotion Recall norepinephrine levels.

SECONDARY OUTCOMES:
Change in high frequency power heart rate variability (hf-HRV) in Ln msec (square) | Up to 4 weeks
  High frequency power heart rate variability (hf-HRV) will be determined by averaging high frequency values for 4-min segments within each phase (Baseline, Emotion Recall), and change will be calculated (Emotion Recall minus Baseline). Data will be collected using a Digital Holter ECG Recorder - 5 Lead, 2 Channel.
Left ventricular ejection fraction (%) | 12 months
  A trans-thoracic echocardiogram will be performed with computation of ejection fraction according to current guidelines.
Average Global Longitudinal Strain (GLS) | 12 months
  Global Longitudinal Strain (GLS) will be assessed using off-line analysis software (TomTec imaging systems). GLS will be calculated as the average left ventricular longitudinal strain across the segments obtained using apical two, three, and four-chamber views. Because myocardial contraction results in left ventricular shortening in systole, GLS is a negative value.

OTHER OUTCOMES:
Proportion of patients with major adverse cardiac and cerebrovascular events | 12 months
  Composite of death from any cause, recurrence of TS, stroke, transient ischemic attack, and myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Salmoirago-Blotcher, MD, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated under the project will be shared as per National Institutes of Health (NIH) Grant Policy and Lifespan Institutional Review Board guidelines. De-identified research data will be made available in a timely manner once the main findings from the final research data set have been accepted for publication. Access to these data will be available for educational or research purposes. Data will be de-identified to avoid linkages to individual research participants and will be free of variables that could lead to deductive disclosure of the identity of individual subjects.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified research data will be made available once the main findings from the final research data set have been accepted for publication.
Access Criteria: Researchers interested in obtaining the de-identified data and associated documentation (e.g. codebook) can make a request to the principal investigator. requestors will be asked to sign a data sharing agreement that includes conditions to 1) protect the identity of participants, 2) limit use of data for educational and research purposes, and 3) prevent transfer of data to other users, and 4) acknowledge the data source. The de-identified data will be shared using Excel or Statistical Package for the Social Sciences (SPSS) file formats.

REFERENCES:
- [Derived] Salmoirago-Blotcher E, Keirns NG, Ouaddi S, Tripolone J, Liu C, Breault C, Dettmer A. Chronic adrenocortical activity and onset of Takotsubo syndrome. Eur J Cardiovasc Nurs. 2026 Jan 21:zvag023. doi: 10.1093/eurjcn/zvag023. Online ahead of print. PMID 41562264